CLINICAL TRIAL: NCT02746211
Title: An Open Label Dose-Ranging Influenza Challenge Study in Healthy Volunteers
Brief Title: Influenza Challenge Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RIS-110 (DEE-CS-002)
Record Dates: First submitted 2016-02-23; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-02

CONDITIONS: Influenza
Keywords: immunology; pathogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Titre Influenza virus (Experimental): High Titre Influenza virus
  Interventions: Biological: High Titre Influenza virus
- Medium - High Influenza virus (Experimental): Medium - High Influenza virus
  Interventions: Biological: Medium - High Influenza virus
- Medium Low Titre Influenza virus (Experimental): Medium Low Titre Influenza virus
  Interventions: Biological: Medium Low Titre Influenza virus
- Low titre Influenza Vaccine (Experimental): Low titre Influenza Vaccine
  Interventions: Biological: Low titre

INTERVENTIONS:
Biological: High Titre Influenza virus — High Titre Influenza virus
  Arms: High Titre Influenza virus
Biological: Medium - High Influenza virus — Medium - High Influenza virus
  Arms: Medium - High Influenza virus
Biological: Medium Low Titre Influenza virus — Medium Low Titre Influenza virus
  Arms: Medium Low Titre Influenza virus
Biological: Low titre — Low titre
  Arms: Low titre Influenza Vaccine

SUMMARY:
A study to determine the infectious titre of an Influenza A (H1N1) (A/New Caledonia/20/99) virus for use in other Influenza challenge studies for the development of Influenza vaccines, antiviral agents and to better understand the host response to Influenza infection.

DETAILED DESCRIPTION:
The primary aim was to determine the infectious titre of an Influenza A (H1N1) (A/New Caledonia/20/99) virus for use in other Influenza challenge studies for the development of Influenza vaccines, antiviral agents and to better understand the host response to Influenza infection.

In addition, the safety of the inoculum, the virus shedding from the nasal mucosa following challenge with Influenza., changes in mRNA and protein expression from blood and nasal brush samples. were assessed Self reported symptoms following challenge were recorded. Samples were taken to facilitate validation of CMI and other immunologically relevant assays in development

Overall Trial Design:

For each group of subjects, quarantine, challenge phase, release from quarantine and decontamination occured concurrently at the designated study site throughout the challenge phase of the study.

The volunteers were be stratified into four groups depending on their intended challenge titre of virus:

High titre Medium-high titre Medium-low titre Low titre Influenza inoculation (nasal drops)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive.
* Comprehension of the study requirements;availability for the required study period, ability to attend scheduled study visits, and willingness to participate in the inpatient challenge.
* Willingness to provide written consent for participation after reading the Consent Form and after having adequate opportunity to discuss the study with an investigator or qualified deputy.
* Good general health status as determined by a screening evaluation no greater than 45 days prior to the quarantine and challenge phase.
* For female subjects, provision of a history of reliable contraceptive practices [hysterectomy or bilateral tubal ligation, oral or implanted contraceptive use, intrauterine device, barrier method plus spermicide, history of a single male partner with vasectomy, or a history of abstinence deemed credible by the investigator(s)]. The provision of this history does NOT replace the requirement to perform, and obtain negative results in, pregnancy tests.

Exclusion Criteria:

* Presence of any significant acute or chronic, uncontrolled medical or psychiatric illness,
* Health care workers (including doctors, nurses, medical students and allied healthcare professionals) anticipated to have patient contact within two weeks of viral challenge. Healthcare workers who volunteer should not work with patients until 14 days after challenge or until their symptoms are fully resolved.
* Venous access deemed inadequate for the phlebotomy demands of the study.
* Positive serologic tests for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
* Evidence of drug abuse or a positive urine Class A drug or alcohol screen.
* Female subjects, who are known to be pregnant or who have a positive urine β-HCG detected prior to challenge.
* Chronic use of any medication or other product (prescription or over-the-counter), for symptoms of rhinitis or nasal congestion or for any chronic nasopharyngeal complaint, or chronic use of any intranasal medication for any indication.
* Any history during adulthood of asthma of any etiology (chronic obstructive pulmonary disease), or any use of a bronchodilator or other asthma medication within adulthood.
* Smokers unwilling/unable to desist for the quarantine phase duration of the study.
* Subject is type I or type II diabetic.
* Subject is allergic to Gentamicin.
* Acute use of any medication or other product, prescription or over-the-counter, for symptoms of rhinitis or nasal congestion within seven (7) days prior to challenge. This includes any corticosteroid or beta agonist containing nasal spray.
* An Abnormal ECG deemed clinically relevant by the Investigator(s).
* Any anatomic or neurologic abnormality impairing the gag reflex or conducive to aspiration, or history suggestive of such a problem or any abnormality significantly altering the anatomy of the nose or nasopharynx.
* Receipt of systemic glucocorticoids (in a dose ≥5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within six months prior to challenge.
* Receipt of any investigational drug within six (6) months prior to challenge, or prior participation in a clinical trial of any Influenza vaccine, or any investigational vaccine or experimental Influenza viral challenge delivered directly to the respiratory tract within 1 year prior to challenge.
* Presence of any febrile illness or symptoms of upper viral respiratory infection:

  1. existing on the day of challenge or between admission for Influenza challenge and administration of the challenge inoculum. (Such subjects may be re-evaluated for enrollment after resolution of the illness);
  2. within two (2) weeks prior to challenge or if challenge is set to occur during November, December, January, February, or March if there are any symptoms suggestive of viral respiratory infection occurring between screening and challenge.
* History of frequent epistaxis (nose bleeds).
* Presence of household member or close contact (for an additional two weeks after discharge from the isolation facility) who is: (a) less than 3 years of age; (b) any person with any known immunodeficiency; (c) any person receiving immunosuppressant medications; (d) any person undergoing or soon to undergo cancer chemotherapy within 28 days of challenge; (e) any person who has diagnosed emphysema or COPD, is elderly residing in a nursing home, or with severe lung disease or medical condition including but not exclusive to the conditions listed in Appendix 8; or (f) any person who has received a transplant (bone marrow or solid organ).
* Any laboratory test which is abnormal and which is deemed by the Investigator(s) to be clinically significant. (This includes blood chemistry, haematology, cardiac iso-enzymes, or urinalysis).
* Known IgA deficiency, immotile cilia syndrome, or Kartagener's syndrome.
* History of seasonal hay fever or a seasonal allergic rhinitis (SAR), including the use of symptomatic prescription only medication and non prescription medication.
* As a result of the medical interview, physical exam, or screening investigations, the Investigator(s) considers the subject unfit for the study.
* Those employed or immediate relatives of those employed at Retroscreen Virology or the study site.
* Receipt of a northern hemisphere seasonal influenza vaccine in the 2006/07/08 winter seasons.
* Receipt of any systemic chemotherapy agent at any time.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The infection rate of an Influenza (A/New Caledonia/20/99) virus. in human volunteers | 14 days

SECONDARY OUTCOMES:
Self Reported Symptoms | 14 days
  Volunteers complete a standardized diary card, rating there symptoms from 0 to 3. The total score for each day is reported.
Virus Shedding from Nasal Mucosa | 14 days
  Nasal wash samples are taken daily and virus titre measured using tissue culture and reported in TCID50.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lambkin-Williams, PhD, Principal Investigator — 020 7756 1300
Locations (1):
- hVIVO Services Ltd, QMB Bioenterprise building, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only in anonymised form